CLINICAL TRIAL: NCT02535091
Title: An Open Label, Multicenter, Safety and Pharmacokinetic Study of YKP3089 as Adjunctive Therapy in Subjects With Partial Onset Seizures
Brief Title: Safety and Pharmacokinetic Study of YKP3089 as Adjunctive Therapy in Subjects With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Life Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YKP3089C021
Record Dates: First submitted 2015-08-21; First posted 2015-08-28 (Estimated); Results first posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-04

CONDITIONS: Partial Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Cenobamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YKP3089 (Experimental): Multiple dose
  Interventions: Drug: YKP3089

INTERVENTIONS:
Drug: YKP3089 — see above
  Other Names: other anti-epileptic drug (AED)

SUMMARY:
This is a multicenter, open label study to assess the safety and pharmacokinetics of YKP3089 as adjunctive therapy in subjects with partial onset seizures. Initially, subjects taking phenytoin or phenobarbital will be enrolled followed by additional subjects taking anti-epileptic drugs (AED) other than phenytoin and phenobarbital to further investigate long-term safety.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria

1. Male or female and greater than or equal to 18 years of age at the time of signing the informed consent. The upper age limit is 70 years inclusive.
2. Weight at least 30 kg
3. Written informed consent signed by the subject or legal guardian prior to entering the study in accordance with the International Conference on Harmonization Good Clinical Practices (ICH GCP) guidelines. If the written informed consent is provided by the legal guardian because the subject is unable to do so, a written or verbal assent from the subject must also be obtained. In Germany, only the subject may sign the informed consent form in accordance with ICH guidelines.
4. A diagnosis of partial epilepsy according to the International League Against Epilepsy's Classification of Epileptic Seizures. Diagnosis should have been established by clinical history and an electroencephalogram (EEG) that is consistent with localization related epilepsy; normal interictal EEGs will be allowed provided that the subject meets the other diagnosis criterion (ie, clinical history).
5. Have uncontrolled partial seizures and require additional AED therapy despite having been treated with at least one AED within approximately the last 2 years.
6. Currently on stable antiepileptic treatment regimen:

   1. Subject must have been receiving stable doses of 1 to 3 AEDs for at least 3 weeks prior to Visit 2
   2. Vagal nerve stimulator (VNS) will not be counted as an AED; however, the parameters must remain stable for at least 4 weeks prior to baseline. The VNS must have been implanted at least 5 months prior to Visit 1.
   3. Benzodiazepines taken at least once per week during the 1 month prior to Visit 1 for epilepsy, or for anxiety or sleep disorder, will be counted as 1 AED and must be continued unchanged throughout the study. Therefore only a maximum of 2 additional approved AEDs will be allowed.
7. Computed tomography (CT) or magnetic resonance imaging (MRI) scan performed within the past 10 years that ruled out a progressive cause of epilepsy. If a CT or MRI has not been performed within the past 10 years, one must be performed prior to randomization.
8. Ability to reach subject by telephone.
9. Use of an acceptable form of birth control by female subjects of childbearing potential

Exclusion Criteria

1. History of any serious drug-induced hypersensitivity reaction (including but not limited to Stevens Johnson syndrome, toxic epidermal necrolysis, drug reaction with eosinophilia and systemic symptoms) or any drug-related rash requiring hospitalization.
2. History of any drug-induced rash or hypersensitivity reaction.
3. History of a first degree relative with a serious cutaneous drug-induced adverse reaction.
4. History of serious systemic disease, including hepatic insufficiency, renal insufficiency, a malignant neoplasm, any disorder in which prognosis for survival is less than 3 months, or any disorder which in the judgment of the investigator will place the subject at excessive risk by participation in a controlled trial
5. Subjects taking phenytoin must not be taking phenobarbital or primidone; subjects taking phenobarbital must not be taking phenytoin or primidone
6. Subjects taking concomitant AEDs other than phenytoin or phenobarbital, must not be taking phenytoin or phenobarbital or primidone
7. Subjects with clinical evidence of phenytoin or phenobarbital toxicity
8. A history of nonepileptic or psychogenic seizures
9. Presence of only nonmotor simple partial seizures or primary generalized epilepsies
10. Presence of Lennox-Gastaut syndrome
11. Scheduled epilepsy surgery within 8 months after Visit 1
12. Subjects implanted with or planning to have implantation of deep brain stimulator
13. Pregnancy or lactation
14. Any clinically significant laboratory abnormality that in the opinion of the investigator would exclude the subject from the study
15. Evidence of significant active hepatic disease. Stable elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) due to concomitant medication(s) will be allowed if they are less than 3 times the upper limit of normal (ULN)
16. An active central nervous system (CNS) infection, demyelinating disease, degenerative neurologic disease, or any CNS disease deemed to be progressive during the course of the study that may confound the interpretation of the study results
17. Any clinically significant psychiatric illness, psychological, or behavioral problems that, in the opinion of the investigator, would interfere with the subject's ability to participate in the study
18. Presence of psychotic disorders and/or unstable recurrent affective disorders evident by use of antipsychotics; presence or recent history (within 6 months) of major depressive episode
19. History of alcoholism, drug abuse, or drug addiction within the past 2 years
20. Current use of felbamate with less than 18 months of continuous exposure
21. Current or recent (within the past year) use of vigabatrin or ezogabine. Subjects with a prior history of treatment with vigabatrin must have documentation showing no evidence of a vigabatrin associated clinically significant abnormality in a visual perimetry test. Subjects with a prior history of treatment with ezogabine should have no evidence of retinal abnormalities with funduscopic features similar to those seen in retinal pigment dystrophies.
22. History of status epilepticus within 3 months of Visit 1
23. Screening laboratory investigation demonstrates abnormal renal function
24. Absolute neutrophil count less than 1500/µL
25. Clinical or ECG evidence of serious cardiac disease, including ischemic heart disease, uncontrolled heart failure, and major arrhythmias, or relevant replicated changes in QT intervals (QTcF less than 340 msec or greater than 450 msec in males and greater than 470 msec in females)
26. Platelet counts lower than 80,000/µL in subjects treated with Valproic acid (divalproex sodium) (VPA)
27. A "yes" answer to Question 1 or 2 of the Columbia Suicide Severity Rating Scale (C-SSRS) (Baseline/Screening version) Ideation Section in the past 6 months or a "yes" answer to any of the Suicidal Behavior Questions in the past 2 years.
28. More than 1 lifetime suicide attempt
29. Participation in any other trials involving an investigational product or device within 30 days of screening (or longer, as required by local regulations)
30. Current use of any of the following medications: clopidogrel, fluvoxamine, amitriptyline, clomipramine, bupropion, methadone, ifosfamide, cyclophosphamide, efavirenz, fosphenytoin, ethotoin, mephenytoin, or natural progesterone (within 1 month of Visit 1)
31. History of positive antibody/antigen test for hepatitis B, hepatitis C, or HIV
32. Presence of congenital short QT syndrome
33. A history of previous exposure to YKP3089

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1345 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kamin, MD, Study Director — SK Life Science, Inc.
Locations (121):
- United States (39):
  - Xen Institute, Phoenix, Arizona
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - Arkansas Epilepsy Program, Little Rock, Arkansas
  - Kaiser Permanente - Southern California Medical Group, Anaheim, California
  - Neuro Pain Medical Center, Fresno, California
  - California Pacific Medical Center, San Francisco, California
  - Blue Sky Neurology, Englewood, Colorado
  - Bradenton Research Center Inc, Bradenton, Florida
  - NW FL Neurology Center, Gulf Breeze, Florida
  - Emory Brain Health Center, Atlanta, Georgia
  - Georgia Neurology and Sleep Medicine Associates, Suwanee, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants In Epilepsy and Neurology PLLC, Boise, Idaho
  - MacFarland Clinic, Ames, Iowa
  - Maine Medical Partners Neurology, Scarborough, Maine
  - The John Hopkins University School of Medicine, Baltimore, Maryland
  - Klein, Pavel (Private Practice), Bethesda, Maryland
  - Neurology Clinic PC, Waldorf, Maryland
  - Minneapolis Clinic of Neurology, Minneapolis, Minnesota
  - Comprehensive Epilepsy Care Center for Children and Adults PC, Chesterfield, Missouri
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - NYU Langone Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Cincinnati, Physicians Company, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Providence Neurological Specialty Clinic, Portland, Oregon
  - Penn Epilepsy Center, Department of Neurology, Philadelphia, Pennsylvania
  - Thomas Jefferson University Comprehensive Epilepsy Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Epilepsy Care Center, Austin, Texas
  - Hunt Regional Medical Partners, Greenville, Texas
  - Baylor Scott and White Research Institute, Temple, Texas
  - University of Virginia, School of Medicine, Charlottesville, Virginia
  - University of Washington School of Medicine, Seattle, Washington
  - UW Medicine, Valley Medical Center, Seattle, Washington
  - Dean and St. Mary's Outpatient Center, Madison, Wisconsin
- Argentina (3):
  - Centro de Educacion Medica e Investigaciones Clinicas (CEMIC), Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hogar de Dia Casa Jesi, Buenos Aires
  - Instituto de Neurociencias de Fundacion Favaloro, Buenos Aires
- Australia (12):
  - Flinders Medical Centre, Bedford Park
  - Eastern Health, Box Hill Hospital, Box Hill
  - Royal Prince Alfred Hospital, Camperdown
  - Strategic Health Evaluators, Chatswood
  - Monash Medical Centre, Clayton
  - St. Vincent's Hospital Melbourne, Fitzroy
  - Austin Health Melbourne Brain Centre, Heidelberg
  - Royal Brisbane & Women's Hospital, Herston
  - Alfred Health - The Alfred Hospital, Melbourne
  - Melbourne Health (The Royal Melbourne Hospital), Parkville
  - Prince of Wales Hospital, Randwick
  - Westmead Hospital, Westmead
- Bulgaria (4):
  - Multiprofile Hospital for Active Treatment Puls AD, Blagoevgrad
  - Multiprofile Hospital for Active Treatment of Neurology and Pschiatry "Sv. Naum" EAD, Sofia
  - First Multiprofile Hospital for Active Treatment- Sofia EAD, Sofia
  - University Multiprofile Hospital for Active Treatment Aleksandrovska EAD, Sofia
- Chile (3):
  - Centro Neuropsicologia LTDA., La Florida, Santiago Metropolitan
  - Complejo Asistencial Dr. Sotero Del Rio, Puente Alto, Santiago Metropolitan
  - Hospital Base Valdivia, Valdivia
- Czechia (3):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Affidea Praha s.r.o., Prague
  - Fakultni nemocnice v Motole, Prague
- Germany (6):
  - Krankenhaus Mara gGmbH - Epilepsiezentrum Bethel, Bielefeld
  - University of Bonn, Department of Epileptology, Bonn
  - Epilepsiezentrum Kork, Kehl
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Universitätsklinikum Münster, Klinik fur Neurologie mit Institut fur Translationale Neurologie-Epileptologie, Münster
- Hungary (3):
  - Országos Klinikai Idegtudományi Intézet, Budapest
  - Debreceni Egyetem Kenezy Gyula Egyetemi Korhaz, Debrecen
  - Bacs Kiskun Megyei Korhaz, Kecskemét
- Mexico (5):
  - Neurociencias Estudios Clinicos S.C., Culiacán
  - Grupo Medico Camino S.C., Mexico City
  - Human Science Research Trials S. de R.L. de C.V., Mexico City
  - Centro de Investigacion Grupo Vitamagen, Monterrey
  - Clinical Research Institute S.C., Tlalnepantla
- Poland (6):
  - Centrum Neurologii Krzysztof Selmaj, Lodz, Lódzkie
  - Centrum Leczenia Padaczki i Migreny, Krakow, Malopolski
  - Fundacja Epileptologii Prof Jerzego Majkowskiego, Warsaw, Masovian Voivodeship
  - Instytut Psychiatrii i Neurologii, Warsaw, Masovian Voivodeship
  - Novo-Med Zielinski i wsp. Sp.J., Katowice, Silesian Voivodeship
  - Copernicus Podmiot Leczniczy Sp. z o.o., Gdansk
- Russia (6):
  - FSBI National Medical Research Centre of Psychiatry and Neurology n.a. V.P. Serbskiy of MoH of RF, Moscow
  - SBHI of Perm Region, Perm Territorial Clinical Hospital, Centre for Multiple Sclerosis, Perm
  - FSBI National Medical Research Centre of Psychiatry and Neurology n.a. V.M. Bekhterev of MoH of RF, Saint Petersburg
  - FSBI of Science, Institute of Human Brain n.a. N.P. Bekhtereva of RAN, Laboratory of Stereotaxic Methods, Saint Petersburg
  - SBHI Samara Regional Clinical Hospital n.a. V.D. Seredavin, Neurology and Neurosurgery Departments, Samara
  - SBGEI of HPE Smolensk State Medical University of MoH of RF, Chair Neurology and Neurosurgery, Smolensk
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Institute of Mental Health, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Kragujevac, Kragujevac
- South Korea (6):
  - Dong-A University Hospital, Busan
  - Keimyung University Dongsan Hospital, Daegu
  - Severance Hospital at Yonsei University Health System, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
- Spain (9):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Parque Tecnológico de la Salud, Granada
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Thailand (2):
  - Faculty of Medicine, Chiang Mai University, Chiang Mai, Muang
  - King Chulalongkorn Memorial Hospital, Faculty of Medicine, Chulalongkorn University, Bangkok, Pathumwan
- Ukraine (9):
  - Municipal Institution Dnipropetrovsk Regional Clinical Hospital, Dnipro
  - Communal Non-Commercial Enterprise of Kharkiv Regional Counsil "Regional clinical psychiatric hospital #3", Kharkiv
  - Kharkiv Railway Clinical Hospital #1 of the Health Center Branch of JSC Ukrzaliznytsia, Kharkiv
  - Communal Noncommercial Enterprise of Lviv Regional Council "Lviv Regional Clinical Hospital", Lviv
  - Municipal Non-Commercial Enterprise Odesa Regional Medical Center for Mental Health of Odessa Regional Council, Odesa
  - Municipal Non-Commercial Enterprise Odesa Regional Medical Center, Odesa
  - Municipal Institution Odesa Regional Psychiatric Hospital #2, Oleksandrivka
  - Municipal Non-Commercial Enterprise "Ternopil Regional Clinical Psychoneurological Hospital" of Ternopil Regional Council, Ternopil
  - Communal Non-profit Enterprise "Vinnytsia Regional Clinical Psycho-Neurological Hospital", Vinnytsia

REFERENCES:
- [Derived] O'Dwyer R, Stern S, Wade CT, Guggilam A, Rosenfeld WE. Safety and Efficacy of Cenobamate for the Treatment of Focal Seizures in Older Patients: Post Hoc Analysis of a Phase III, Multicenter, Open-Label Study. Drugs Aging. 2024 Mar;41(3):251-260. doi: 10.1007/s40266-024-01102-3. Epub 2024 Mar 6. PMID 38446341
- [Derived] Sperling MR, Abou-Khalil B, Aboumatar S, Bhatia P, Biton V, Klein P, Krauss GL, Vossler DG, Wechsler R, Ferrari L, Grall M, Rosenfeld WE. Efficacy of cenobamate for uncontrolled focal seizures: Post hoc analysis of a Phase 3, multicenter, open-label study. Epilepsia. 2021 Dec;62(12):3005-3015. doi: 10.1111/epi.17091. Epub 2021 Oct 11. PMID 34633084

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Discrepancies can be found in the Protocol Enrollment number and the Participant Flow data. This discrepancy can be explained by the understanding that the Protocol Enrollment number refers to all participants that signed an informed consent form, while the Participant Flow data only takes into account participants that were dosed with at least one dose of study drug.
Groups:
- YKP3089 and Phenytoin: Subjects taking phenytoin and cenobamate.
- YKP3089 and Phenobarbital: Subjects taking phenobarbital and cenobamate.
- YKP3089 and Other AEDs: Subjects taking AEDs other than phenobarbital and phenytoin and taking cenobamate.
Period: Overall Study
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs
Started | 83 | 37 | 1220
Completed | 22 | 5 | 236
Not Completed | 61 | 32 | 984
Not completed — Entered Expanded Access Program (EAP)/Navigator | 34 | 18 | 575
Not completed — Withdrawal by Subject | 14 | 5 | 121
Not completed — Adverse Event | 9 | 4 | 170
Not completed — Other | 4 | 3 | 81
Not completed — Lost to Follow-up | 0 | 1 | 19
Not completed — Protocol Violation | 0 | 1 | 11
Not completed — Pregnancy | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs | Total
Number analyzed (Participants) | 83 | 37 | 1220 | 1340
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 76 | 35 | 1187 | 1298
  >=65 years | 7 | 2 | 33 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 15 | 624 | 667
  Male | 55 | 22 | 596 | 673
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 0 | 50 | 59
  Asian | 2 | 6 | 65 | 73
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 5 | 6
  Black or African American | 4 | 1 | 42 | 47
  White | 46 | 28 | 991 | 1065
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 21 | 2 | 67 | 90
Height [Mean (Standard Deviation); unit: cm] | 170.42 (11.365) | 167.92 (10.064) | 169.31 (10.257) | 169.34 (10.322)
Weight [Mean (Standard Deviation); unit: kg] | 80.82 (21.489) | 75.91 (16.882) | 77.11 (18.442) | 77.30 (18.612)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.69 (6.126) | 26.78 (5.280) | 26.87 (5.993) | 26.92 (5.982)

OUTCOME MEASURES:

1. Primary Outcome: Summary of Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as Adverse events (AEs) with onset on or after the start of study medication, up to last dose date of study medication + 14 days or onset before study medication and worsened after starting study medication, up to last dose date of study medication + 14 days.
Time Frame: 1 day to up to 215 weeks after first dose.
Measure: Number; unit: participants
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs
Number analyzed (Participants) | 83 | 37 | 1220
participants
  At least 1 TEAE | 76 | 35 | 1104
  At least 1 treatment-related TEAE | 57 | 29 | 923
  TEAE with outcome of death | 1 | 0 | 5
  TEAE leading to study drug discontinuation | 9 | 6 | 168
  At least 1 serious TEAE | 15 | 6 | 217
  At least 1 severe TEAE | 10 | 4 | 148

2. Other Pre Specified Outcome: Vital Signs: Meeting Abnormal Criteria (Post-Baseline Measurement)
Description: Subjects with At Least 1 Post-Baseline Measurement Meeting Abnormal Criteria. Changes in systolic and diastolic blood pressure, pulse rate, respiratory rate, temperature, weight, and height in each safety evaluable group were small and not clinically meaningful.
Time Frame: 1 day to up to 215 weeks after first dose.
Measure: Number; unit: participants
Groups:
- Safety Population: All subjects enrolled in the study who received at least 1 dose of study drug medication were considered safety evaluable subjects.
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs | Safety Population
Number analyzed (Participants) | 83 | 37 | 1220 | 1340
participants
  Systolic blood pressure <90 mmHg | 3 | 3 | 58 | 64
  Systolic blood pressure >140 mmHg | 26 | 15 | 310 | 351
  Systolic blood pressure >160 mmHg | 7 | 0 | 44 | 51
  Diastolic blood pressure <50 mmHg | 0 | 2 | 41 | 43
  Diastolic blood pressure >90 mmHg | 29 | 12 | 318 | 359
  Diastolic blood pressure >100 mmHg | 7 | 2 | 68 | 77
  Pulse rate <60 bpm | 35 | 14 | 446 | 495
  Pulse rate >100 bpm | 2 | 1 | 79 | 82
  Body weight: Decrease of ≥7% from baseline | 21 | 12 | 373 | 406
  Body weight: Increase of ≥7% from baseline | 19 | 5 | 272 | 296
  Respiratory rate <12 breaths/min | 2 | 2 | 33 | 37
  Respiratory rate >20 breaths/min | 22 | 6 | 247 | 275
  Temperature >38.0°C | 0 | 1 | 5 | 6
  Temperature <36.0°C | 33 | 12 | 384 | 429

3. Other Pre Specified Outcome: Exposure to Study Dose - Length (Weeks)
Description: Exposure to Study Dose was measured in Safety Population. Modal daily dose defined as the dose taken the most days during the reporting phase or study; in case of ties, modal dose was defined as the highest dose level between the two doses in the tie.
Time Frame: 1 day to up to 215 weeks after first dose.
Measure: Mean (Standard Deviation); unit: weeks/months/mg
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs | Safety Population
Number analyzed (Participants) | 83 | 37 | 1220 | 1340
weeks/months/mg
  Length of Exposure (Weeks) - Overall | 123.96 (62.885) | 119.48 (81.612) | 129.28 (65.436) | 128.68 (65.753)
  Length of Exposure (Weeks) - Maintenance Phase | 122.4 (21.89) | 136.7 (61.93) | 131.6 (50.33) | 131.2 (50.75)

4. Other Pre Specified Outcome: YKP3089 Plasma Levels (mcg/mL)
Description: At Visit 8 and Visit 9, 2 blood samples were collected for the determination of YKP3089 plasma levels (YKP3089 and concomitant AED doses must have been stable for 2 weeks prior to these visits), at arrival and 30 minutes to 4 hours after the most recent dose.
  Plasma levels of phenytoin and phenobarbital were stable during the titration. The endpoint values are based on pharmacokinetic (PK) population.
Time Frame: Day 85 and Day 99 after first dose.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs
Number analyzed (Participants) | 83 | 37 | 364
mcg/mL
  Visit 8 (Day 85) / Arrival at clinic | 12.5051 (5.80730) | 12.4071 (4.71288) | 14.6904 (5.99973)
  Visit 8 (Day 85) / Post-Dose | 13.7470 (6.02498) | 14.6900 (4.44020) | 15.8694 (5.92152)
  Visit 9 (Day 99) / Arrival at clinic | 11.8173 (5.36440) | 13.2607 (5.46875) | 15.4764 (5.94161)
  Visit 9 (Day 99) / Post-Dose | 13.4618 (5.69905) | 15.0770 (5.25885) | 16.4892 (5.87959)

5. Other Pre Specified Outcome: Exposure to Study Dose - Length (Months)
Description: as for outcome 3
Time Frame: 1 day to up to 215 weeks after first dose.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs | Safety Population
Number analyzed (Participants) | 83 | 37 | 1220 | 1340
months
  Length of Exposure (Months) - Overall | 28.543 (14.4801) | 27.512 (18.7922) | 29.768 (15.0675) | 29.630 (15.1404)
  Length of Exposure (Months) - Maintenance Phase | 28.18 (11.949) | 31.47 (14.261) | 30.31 (11.589) | 30.20 (11.686)

6. Other Pre Specified Outcome: Average Exposure to Study Dose
Description: as for outcome 3
Time Frame: 1 day to up to 215 weeks after first dose.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs | Safety Population
Number analyzed (Participants) | 83 | 37 | 1220 | 1340
mg
  Modal Daily Dose (mg) - Overall | 223.34 (100.528) | 183.11 (105.500) | 219.32 (107.154) | 218.57 (106.808)
  Modal Daily Dose (mg) - Maintenance Phase | 244.7 (82.84) | 222.4 (85.13) | 244.5 (88.32) | 244.0 (87.91)

ADVERSE EVENTS:
Time Frame: Adverse event data is collected from the initiation of any study procedures (Visit 1) to the end of treatment follow-up. The time frame of each participant varies from 1 day to up to 215 weeks on study treatment. The AE reporting period is defined as 30 days following the last administration of study treatment for serious adverse events (SAEs) and 14 days following the last administration of study treatment for all other AEs.
Arm/Group | YKP3089 and Phenytoin | YKP3089 and Phenobarbital | YKP3089 and Other AEDs
All-Cause Mortality (participants affected / at risk) | 2/83 | 0/37 | 8/1220
Serious Adverse Events (participants affected / at risk) | 15/83 | 6/37 | 217/1220
Other Adverse Events (participants affected / at risk) | 76/83 | 35/37 | 1104/1220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | YKP3089 and Phenytoin (N=83) | YKP3089 and Phenobarbital (N=37) | YKP3089 and Other AEDs (N=1220)
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 7
Corona virus infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis bacterial (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 4
Ankle fracture (Infections and infestations) | 0 | 1 | 2
Fall (Infections and infestations) | 0 | 1 | 5
Intentional overdose (Infections and infestations) | 1 | 0 | 1
Toxicity to various agents (Infections and infestations) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 6
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 6
Dizziness (Nervous system disorders) | 0 | 0 | 5
Epilepsy (Nervous system disorders) | 0 | 0 | 8
Generalized tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 2
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 0 | 0
Postictal paralysis (Nervous system disorders) | 0 | 0 | 6
Postictal state (Nervous system disorders) | 0 | 0 | 4
Seizure (Nervous system disorders) | 1 | 1 | 27
Seizure cluster (Nervous system disorders) | 0 | 1 | 2
Status epilepticus (Nervous system disorders) | 0 | 0 | 7
Anger (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 5
Suicide attempt (Psychiatric disorders) | 1 | 0 | 4
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6
Arterial haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 2
Hopitalisation (Surgical and medical procedures) | 0 | 0 | 1
Neurolysis (Surgical and medical procedures) | 0 | 0 | 1
Vagal nerve stimulator implantation (Surgical and medical procedures) | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gliosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Sarcoidosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 3
Complications associated with device (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Pelvic mass (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Serositis (General disorders) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 0 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 2
Mental status changes (Psychiatric disorders) | 0 | 0 | 3
Mood disorder due to a general medical condition (Psychiatric disorders) | 0 | 0 | 1
Postictal psychosis (Psychiatric disorders) | 0 | 0 | 1
Psychogenic seizure (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 3
Schizophrenia (Psychiatric disorders) | 0 | 0 | 1
Substance use disorder (Psychiatric disorders) | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 2
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 2
Pelvic haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 2
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 3
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fibrin D dimer increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Cortical dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 1
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 2
Cerebral atrophy (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 2
Focal dyscognitive seizures (Nervous system disorders) | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 2
Migraine (Nervous system disorders) | 0 | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Poor sucking reflex (Nervous system disorders) | 0 | 0 | 1
Post-traumatic epilepsy (Nervous system disorders) | 0 | 0 | 2
Presyncope (Nervous system disorders) | 0 | 0 | 1
Radial nerve palsy (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 3
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Vertebral artery dissection (Nervous system disorders) | 0 | 0 | 1
Wernicke's encephalopathy (Nervous system disorders) | 0 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 2
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Adrenal mass (Endocrine disorders) | 0 | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Tetany (Metabolism and nutrition disorders) | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
Abscess oral (Infections and infestations) | 0 | 0 | 1
Appendiceal abscess (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 2
Dengue fever (Infections and infestations) | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 1
Sepsis neonatal (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 2
Vestibular neuronitis (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | YKP3089 and Phenytoin (N=83) | YKP3089 and Phenobarbital (N=37) | YKP3089 and Other AEDs (N=1220)
Diplopia (Eye disorders) | 6 | 2 | 83
Vision blurred (Eye disorders) | 4 | 3 | 48
Nausea (Gastrointestinal disorders) | 5 | 1 | 54
Fatigue (General disorders) | 18 | 8 | 211
Gait disturbance (General disorders) | 6 | 3 | 52
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 23
Ataxia (Nervous system disorders) | 5 | 4 | 49
Balance disorder (Nervous system disorders) | 10 | 3 | 69
Dysarthria (Nervous system disorders) | 1 | 3 | 32
Headache (Nervous system disorders) | 4 | 3 | 115
Nystagmus (Nervous system disorders) | 7 | 1 | 26
Somnolence (Nervous system disorders) | 19 | 15 | 359

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT02535091/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT02535091/SAP_001.pdf